CLINICAL TRIAL: NCT03353324
Title: Comparison of Therapeutic Effects Between Intravitreal Injection of Bevacizumab With Intravitreal Injection of Bevacizumab and Targeted Laser Photocoagulation of Non Perfused Areas of Retina in Patients With Acute Retinal Vein Occlusion
Acronym: bevacizumab
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9696
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2017-05

CONDITIONS: Retinal Vein Occlusion With Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravitreal injection of bevacizumab (Active Comparator)
  Interventions: Drug: intravitreal injection of bevacizumab
- intravitreal injection of bevacizumab+ targeted laser (Active Comparator): Intervention intravitreal bevacizumab injection + targeted laser photocoagulation of retinal non perfused areas
  Interventions: Radiation: intravitreal injection of bevacizumab+ targeted laser

INTERVENTIONS:
Drug: intravitreal injection of bevacizumab — under gone 3 intravitreal injection of bevacizumab monthly and examine monthly for Visual acuity and central macular thickness, if in month four or more the CMT is more than 250 micrometer and the visual acuity is less than 8/10 the injection is repeatet and follow up in this manner is continued until 9 months.
  Arms: intravitreal injection of bevacizumab
Radiation: intravitreal injection of bevacizumab+ targeted laser — patients in this group undergone laser photocoagulation of retinal non perfused areas based on FAG wide field imaging .
  After 9 month follow up the outcomes such as Vusal acuity, Central macular thickness, intraocular pressure, neovascular formation are compared
  Arms: intravitreal injection of bevacizumab+ targeted laser

SUMMARY:
Patients with new onset retinal vein occlusion in less than 3 month whom has visual acuity less than 20/40 and central macular thickness more than 250micrometer and non perfused areas of retina more than 10 DD are included in over study and devided into 2 groups randomizely, Group A under gone 3 intravitreal injection of bevacizumab monthly and examine monthly for Visual acuity and central macular thickness, if in month four or more the CMT is more than 250 micrometer and the visual acuity is less than 8/10 the injection is repeated and follow up in this manner is continued until 9 months.

Group B is as the same of group A but patients in this group undergone laser photocoagulation of retinal non perfused areas based on FAG wide field imaging .

After 9 month follow up the outcomes such as Vusal acuity, Central macular thickness, intraocular pressure, neovascular formation are compared,

ELIGIBILITY:
Inclusion Criteria:

* Center-involved macular edema secondary to RVO on clinical exam
* Symptoms less than 3 months
* BCVA= 20/40 or worse
* Mean center point thickness >250 μm
* Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs

One eye per participant is enrolled in the trial

Exclusion Criteria:

* Macular edema due to a cause other than CRVO
* An ocular condition such that visual acuity would not improve from resolution of the edema (eg, foveal atrophy)
* Substantial cataract estimated to have reduced visual acuity by >3 lines
* Prior treatment with intravitreal or peribulbar steroid injection
* History of macular photocoagulation or PRP
* Prior pars plana vitrectomy
* Hx of Intraocular surgery (including cataract extraction)
* uveitis, NVG, exudative AMD, diabetic retinopathy, any malignancy, optic neuropathy, amblyopia
* vitreomacular traction or epiretinal membrane *uncontrolled glaucoma ( > 30mmHg with anti-glaucoma medications)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Every month
  Snellen chart

SECONDARY OUTCOMES:
macular thickness | every month
  OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided